CLINICAL TRIAL: NCT00507676
Title: Lung Function and Structure in Healthy Infants and Infants With Recurrent Wheezing
Status: Completed | Type: Observational
Sponsor: Indiana University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Robert S. Tepper, MD, Phd, Indiana University
Organization: Indiana University (Other)
Other Study IDs: 9909-30
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2011-01

CONDITIONS: Asthma; Wheezing; Infant
Keywords: Asthma; Wheezing; Infant
MeSH Terms: conditions — Asthma; Respiratory Sounds

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We collect hair samples to analyzed for nicotine and cotinine.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group 1: One hundred and sixty healthy infants between 1 and 24 months of age will be evaluated. Subjects will be recruited so that there are 40 subjects within each of four subgroups: 1) Negative ETS exposure and Negative Fm Asthma, 2) Positive ETS exposure and Negative Fm Asthma, 3) Negative ETS exposure and Positive Fm Asthma and 4) Positive ETS exposure and Positive Fm Asthma. Equal numbers of males and females will be recruited. The ethnic composition will be approximately 80% Caucasian and 20% African-American in each of the four groups, which represents the distribution within the cities where infants will be evaluated. Subjects will be excluded if they were born prematurely (<37 weeks gestation), have a history of congenital cardio-respiratory disease, or have history of lower respiratory illness.
- Group 2: Eighty infants between 1 and 24 months of age scheduled for CT scans of the abdomen or chest will be evaluated. Subjects will be excluded if they are born prematurely (<37 weeks gestation), have history of congenital cardio-respiratory disease, or have history of recurrent wheezing.
- Group 3: Eighty infants with recurrent wheezing between 1 and 24 months of age will be evaluated when they are not acutely symptomatic for at least 3 weeks. Subjects will be recruited so that there are 20 subjects within each of four subgroups: 1) Negative ETS exposure and Negative Fm Asthma, 2) Positive ETS exposure and Negative Fm Asthma, 3) Negative ETS exposure and Positive Fm Asthma and 4) Positive ETS exposure and Positive Fm Asthma. Equal numbers of males and females will be recruited. Subjects will be excluded if they were born prematurely (<37 weeks gestation) or have history of congenital cardio -respiratory disease.

SUMMARY:
Infants will be enrolled into this study in one of three groups. First, there will be a group of full term infants with no history of wheezing. Second, there will be a group of infants receiving a ct scan that is non-respiratory related. Third, there will be a group of infants that are born full term but have a history of wheezing of at least 3 episodes. The three groups will be compared to see if there is a difference in lung function, lung structure and lung size. Besides comparing the testing results we will be evaluating environmental and inherited characteristics. There are 2 purposes of this study. The first purpose is: To determine whether asymptomatic groups of infants at high risk for wheezing (Environmental tobacco smoke (ETS) exposure, Fm Asthma, male Gender) have fixed or reversible airway narrowing. The second purpose of this study is: To determine the relative contributions of fixed and reversible airway narrowing in infants with recurrent symptomatic wheezing, and to determine whether fixed and reversible airway narrowing is related to ETS exposure, Fm Asthma, and male Gender.

DETAILED DESCRIPTION:
Among asymptomatic healthy infants decreased airway function is found in infants exposed to environmental tobacco smoke (ETS) or with history of family asthma (Fm Asthma), or male gender. These infants are at significantly greater risk of wheezing during infancy. These findings indicate that genetic and environmental factors affect the mechanical determinants of airway function and that among healthy infants variations of these mechanical determinants contribute to the increased risk of developing airway obstruction severe enough to result in clinical symptoms of wheezing. The mechanisms of reduced airway function in these at risk infants are not known. In adults reduced airway function is a result of airway narrowing, increased airway compliance, or decreased pulmonary elastic recoil. The same is thought to be true in infants. The cause of airway narrowing may be functional (reversible by bronchodilators) or structural (fixed, not reversible by bronchodilators) or have components of both. Fixed determinants of airway narrowing include small absolute airway size, thickened airway wall, decreased elastic recoil, and small airway size relative to lung volume. Reversible determinants include airway hyper-responsiveness and inflammation. Understanding the alterations of airway function that increase the risk of airway disease will be decisive in the development of strategies for the prevention and treatment of wheezing in infants and children, and hence, a reduction of morbidity and mortality.

It is not known whether infants with recurrent wheezing have persistent airway narrowing when not acutely symptomatic, and whether airway function in these infants is related to ETS exposure, Fm Asthma, and male gender. When recurrently wheezy infants are asymptomatic, airway function may be low or normal, and low airway function may be fixed or reversible with a bronchodilator. It is important to determine whether these infants have functional and structural abnormalities when they are not acutely symptomatic, and to determine how lung structure relates to lung function. Only then can we design effective therapeutic interventions for recurrently symptomatic infants, as well as, design early intervention strategies.

The Specific aims of this project are:

Specific Aim # 1: To determine whether asymptomatic groups of infants at high risk for wheezing (Environmental tobacco smoke (ETS) exposure, Fm Asthma, male Gender) have fixed or reversible airway narrowing.

Specific Aim # 2: To determine the relative contributions of fixed and reversible airway narrowing in infants with recurrent symptomatic wheezing, and to determine whether fixed and reversible airway narrowing is related to ETS exposure, Fm Asthma, and male Gender.

We propose to answer these important questions of lung function and structure in infants using state of the art methodologies

ELIGIBILITY:
Inclusion Criteria:

* For all 3 groups in the study

  a) Full term >37 weeks
* Group 2

  a) Must have a CT scan nonrespiratory related
* Group 3 a) Must have had at lease 3 episodes of wheezing

Exclusion Criteria:

* Group 1 and 2

  1. cardio-respiratory disease
  2. history of recurrent wheezing or lower respiratory infections
* Group 3 a) cardio-respiratory disease

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We are recruiting infants with asthma and wheezing from pulmonary outpatient clinics at Riley Hospital for children. The full term healthy infants were recruited by advertisements in the local Indy's Child Magazine. These children were volunteers from Indianapolis and surrounding counties.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2000-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Tepper, MD, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States